CLINICAL TRIAL: NCT06322004
Title: Video-Interpreting in Prehospital Emergency Medicine - Feasibility Study
Status: Recruiting | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Christina Hafner, Principal Investigator, Medical University of Vienna
Other Study IDs: 1718/2022
Record Dates: First submitted 2023-10-25; First posted 2024-03-20 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Communication Barriers
Keywords: Communication barriers; Prehospital emergency medicine; Emergency medicine; Emergency physician

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
50 responsive patients with language barriers will be included in this study. The prehospital emergency physician will start video-interpreting via a tablet. Feasibility, quality of communication, usability as well as changes in diagnosis and treatment will be gathered and analysed.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, at least 18 years old
* awake, responsive patients
* language barrier (Albanian, Dari, Romanian, Turkish, Modern Standard Arabic, Arabic, Farsi, Russian, Hungarian, Bosnian-Croatian-Serbian, Kurdish (Kurmanci), Slovakian, Bulgarian, Polish, and Czech)

Exclusion Criteria:

* unconscious patients
* out-of-hospital cardiac arrest patients
* delay of treatment or transportation due to e-interpreting
* refusal of video-interpreting by the patient

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 50 responsive patients treated by prehospital emergency doctors of the Department of Anaesthesia, Intensive Care and Pain Management (Medical University of Vienna/ General Hospital of Vienna) with language barrier (14 languages Albanian, Dari, Romanian, Turkish, Modern Standard Arabic, Arabic, Farsi, Russian, Hungarian, Bosnian-Croatian-Serbian, Kurdish (Kurmanci), Slovakian, Bulgarian, Polish, and Czech) will be included regarding inclusion and exclusion criteria mentioned above.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-02-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Technical Feasibility | Immediately after use of video-interpreting
  The technical feasibility endpoint evaluates the possibility of video-interpreting.
  The occurrence of technical problems will be reported.
Usability of video-interpreting | Immediately after use of video-interpreting
  The usability will be evaluated after the rescue mission by the prehospital emergency doctor using a questionnaire including following items on a 7-point Likert scale (strongly disagree to strongly agree):
  * Video-translation was easy to use.
  * I feel comfortable to use video-translation during the situation.
  * The amount of time involved to use video-translation has been fitting for me.
  * I would use video-translation again.
  * Video-translation was useful for my healthcare practice in this situation.
Impact on emergency physician's decisions | Immediately after use of video-interpreting
  The impact of video-translation will be evaluated regarding alteration of medical history, treatment or target hospital.

SECONDARY OUTCOMES:
Demographic parameters | Immediately after use of video-interpreting
  Following characteristics of the patients will be recorded:
  Age, Gender, primary diagnosis of the prehospital emergency physician

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No